CLINICAL TRIAL: NCT06090734
Title: Development and Evaluation of 'My Voice': a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Collaborators: Changi General Hospital (Other); Singapore General Hospital (Other); Sengkang General Hospital (Other); National Heart Centre Singapore (Other); Khoo Teck Puat Hospital (Other)
Responsible Party: Principal Investigator, Chetna Malhotra, Associate Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2022/2482
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-02

CONDITIONS: Advance Care Planning; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- My Voice (Experimental): Intervention arm patients will complete the patient version of 'My Voice' at least once every 3 months for 1 year or until they pass away (whichever is earlier).
  Caregivers of patients in the intervention arm will complete the caregiver version of 'My Voice' at least once every 3 months for 1 year (or until the patient passes away, whichever is earlier).
  Interventions: Other: My Voice
- Control (No Intervention): Control arm patients and caregivers will receive usual care.

INTERVENTIONS:
Other: My Voice — The web intervention educates patients about their illness and supports them to make their own Advance Care Planning decisions, update these decisions frequently as their clinical condition changes, and to make the ACP process easier and more accessible. The intervention aims to shift implementation of ACP from a provider-led one-time model to a patient-led dynamic model.
  Arms: My Voice

SUMMARY:
The study aims to develop and evaluate a web-based interactive platform (called 'My Voice') that helps to educate patients with heart failure and their caregivers about heart failure, identify their goals for end-of-life care, and share these with their caregivers and doctors.

DETAILED DESCRIPTION:
The research study consists of 3 phases:

1. Usability testing - to assess the usability of 'My Voice' with patients with heart failure, their caregivers and healthcare providers,
2. Pilot testing - to test the feasibility of implementation and workflow of 'My Voice' and the survey questionnaires with a small group of participants and,
3. Randomized controlled trial- to evaluate the effectiveness of 'My Voice' with a control group who do not receive the intervention in improving patient outcomes

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria for patients are

1. Age ≥ 21 years old
2. Singaporean or Permanent Resident
3. Diagnosed with heart failure
4. Symptoms classified under NYHA class II (with an ejection fraction of less than or equal to 35%), III or IV
5. Intact cognition determined through the Abbreviated Mental Test (AMT) (for pilot testing and main RCT)
6. Ability to speak and read English, Mandarin or Malay
7. Willing to complete a web intervention
8. Easily contactable via mobile phone or landline
9. Have a permanent address in Singapore for at least the next 1 year
10. Not recruited in a previous phase of the study

The inclusion criteria for caregivers are

1. Age ≥ 21 years old
2. Nominated as a healthcare spokesperson by the patient or the main decision maker for the patient (for intervention arm only)
3. Ability to speak and read English, Mandarin or Malay
4. Willing to complete a web intervention
5. Easily contactable via mobile phone or landline
6. Have a permanent address in Singapore for at least the next 1 year

Exclusion criteria for caregivers are:

a) domestic helper

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-03-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who have ACP discussions with their treating doctor at least once during the study period | 1 year from data collection
  will be assessed from medical records and survey
Proportion of patients who have ACP discussions with their caregivers | 1 year from data collection
  will be assessed from the survey
Proportion of patients who prefer life-extending treatments | 1 year from data collection
  will be assessed from the survey

SECONDARY OUTCOMES:
Proportion of patients with psychological distress | 1 year from data collection
  will be assessed from the survey
Peace and acceptance scores | 1 year from data collection
  will be assessed from the survey
Proportion of patients having decision maker | 1 year from data collection
  will be assessed from the survey

CONTACTS AND LOCATIONS:
Overall Officials: Chetna Malhotra, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No